CLINICAL TRIAL: NCT00369824
Title: A Randomized, Open Study to Evaluate the Safety and Immunogenicity of GlaxoSmithKline Biologicals' HPV Vaccine Co-administered Intramuscularly With Boostrix® and/or Menactra™ in Healthy Female Subjects Aged 11-18 Years
Brief Title: Evaluation of Safety and Immunogenicity of Co-administering HPV Vaccine With Other Vaccines in Healthy Female Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 107682
Record Dates: First submitted 2006-08-28; First posted 2006-08-29 (Estimated); Results first posted 2009-10-08 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2016-11

CONDITIONS: Infections, Papillomavirus
Keywords: HPV; HPV, diptheria, pertussis, tetanus, meningitis
MeSH Terms: conditions — Papillomavirus Infections; Whooping Cough; Tetanus; Meningitis

ARMS (6):
- Cervarix + Boostrix/Menactra Group (Experimental): Subjects received Cervarix and Boostrix at Month 0, Menactra and Cervarix at Month 1 and Cervarix alone at Month 6.
  Interventions: Biological: Different formulations of GSK Biologicals' HPV vaccine (580299); Biological: Menactra TM; Biological: Boostrix TM
- Cervarix + Menactra/Boostrix Group (Experimental): Subjects received Menactra and Cervarix at Month 0, Boostrix and Cervarix at Month 1 and Cervarix alone at Month 6.
  Interventions: Biological: Different formulations of GSK Biologicals' HPV vaccine (580299); Biological: Menactra TM; Biological: Boostrix TM
- Cervarix + Boostrix + Menactra Group (Experimental): Subjects received Boostrix, Menactra and Cervarix at Month 0 and Cervarix alone at Months 1 and 6.
  Interventions: Biological: Different formulations of GSK Biologicals' HPV vaccine (580299); Biological: Menactra TM; Biological: Boostrix TM
- Boostrix/Cervarix Group (Experimental): Subjects received Boostrix at Month 0 and Cervarix at Months 1, 2 and 7.
  Interventions: Biological: Different formulations of GSK Biologicals' HPV vaccine (580299); Biological: Menactra TM; Biological: Boostrix TM
- Menactra/Cervarix Group (Experimental): Subjects received Menactra at Month 0 and Cervarix at Months 1, 2 and 7.
  Interventions: Biological: Different formulations of GSK Biologicals' HPV vaccine (580299); Biological: Menactra TM
- Cervarix Group (Experimental): Subjects received Cervarix at Months 0, 1 and 6.
  Interventions: Biological: Different formulations of GSK Biologicals' HPV vaccine (580299)

INTERVENTIONS:
Biological: Different formulations of GSK Biologicals' HPV vaccine (580299) — Three doses of vaccine administered intramuscularly, with the second and third dose given one month and six months after the first dose respectively
Biological: Menactra TM — One dose of vaccine administered intramuscularly
  Arms: Boostrix/Cervarix Group; Cervarix + Boostrix + Menactra Group; Cervarix + Boostrix/Menactra Group; Cervarix + Menactra/Boostrix Group; Menactra/Cervarix Group
Biological: Boostrix TM — One dose of vaccine administered intramuscularly
  Arms: Boostrix/Cervarix Group; Cervarix + Boostrix + Menactra Group; Cervarix + Boostrix/Menactra Group; Cervarix + Menactra/Boostrix Group

SUMMARY:
Infection with human papillomavirus (HPV) has been clearly established as the central cause of cervical cancer. Vaccination of pre-teens and adolescents, ideally before sexual debut and thus before exposure to oncogenic HPV, is a rational strategy for prevention of cervical cancer, and so HPV vaccination could complement the existing pre-adolescent/adolescents platform. Therefore, this Phase 3b study is designed to evaluate the safety and immunogenicity of co-administering Boostrix and/or Menactra with GSK Biologicals' HPV vaccine (580299) as compared to the administration of any of the vaccines alone.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can, and will, comply with the requirements of the protocol should be enrolled in the study.
* A female between, and including, 11 and 18 years of age at the time of the first vaccination.
* Written informed consent obtained from parents/legally acceptable representative of the subject and written informed assent obtained from the subject if the subject is less than 18 years of age, or written informed consent obtained from the subject if the subject is 18 years of age.
* Healthy subjects, as established by medical history and history-directed physical examination, before entering into the study.
* Previously completed routine childhood vaccinations against diphtheria, tetanus and pertussis diseases, according to the recommended vaccination schedule at the time.
* Subjects must have a negative urine pregnancy test.
* Subjects of childbearing potential at the time of study entry are required to be abstinent or use adequate contraceptive precautions for 30 days prior to vaccination. Subjects also are required to agree to continue such precautions for two months after completion of the vaccination series. Female subjects who reach menarche (began menstruating) during the study and therefore become of child-bearing potential are required to agree to follow the same precautions.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period (up to the Month 12/13 visit), in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before and 30 days after each dose of vaccine. Administration of routine vaccines up to 8 days before the first dose of study vaccine is allowed. Enrolment will be deferred until the subject is outside of specified window.
* A woman planning to become pregnant, likely to become pregnant or planning to discontinue contraceptive precautions during the study period and up to two months after the last vaccine dose.
* Pregnant or breastfeeding women.
* Previous vaccination against HPV, or planned administration of any HPV vaccine other than that foreseen by the study protocol during the study period.
* previous administration of components of the investigational vaccine
* Administration of a pre-school booster of diphtheria, tetanus, pertussis vaccine within the previous five years.
* Administration of a diphtheria-tetanus booster or tetanus-diphteria-acellular pertussis (Tdap) vaccine within the previous five years.
* Previous vaccination against Neisseria meningitidis.
* Hypersensitivity to latex.
* Cancer or autoimmune disease under treatment.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine or following any other tetanus toxoid, diphtheria toxoid or pertussis-containing vaccine.
* History of encephalopathy within seven days of administration of a previous dose of pertussis vaccine that is not attributable to another identifiable cause.
* Progressive neurologic disorder, uncontrolled epilepsy or progressive encephalopathy.
* Temperature of >= 105°F within 48 hours of receipt of a prior dose of diphteria- tetanu-pertussis (DTP) vaccine, not due to another identifiable cause.
* Collapse or shock-like state within 48 hours of receipt of a prior dose of DTP vaccine.
* Seizures with or without fever within three days of a prior dose of DTP vaccine.
* Severe Arthus-type hypersensitivity reactions following a prior dose of tetanus toxoid within the previous 10 years.
* Previous history of Guillain-Barré syndrome.
* Any confirmed or suspected immunosuppressive or immunodeficient condition
* Acute disease at the time of enrolment. All vaccines can be administered to persons with a minor illness
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.

Ages: 11 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1330 (Actual)
Dates: Start 2006-09-26; Primary Completion 2007-11-22 (Actual); Study Completion 2008-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (49):
- United States (49):
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Madera, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, Centennial, Colorado
  - GSK Investigational Site, Golden, Colorado
  - GSK Investigational Site, Thornton, Colorado
  - GSK Investigational Site, Cocoa Beach, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Arkansas City, Kansas
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Bossier City, Louisiana
  - GSK Investigational Site, Milford, Massachusetts
  - GSK Investigational Site, Niles, Michigan
  - GSK Investigational Site, Stevensville, Michigan
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Edison, New Jersey
  - GSK Investigational Site, Whitehouse Station, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Cary, North Carolina
  - GSK Investigational Site, Laurinburg, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Sylva, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Boardman, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Greenville, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Uniontown, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Gray, Tennessee
  - GSK Investigational Site, San Angelo, Texas
  - GSK Investigational Site, Burke, Virginia
  - GSK Investigational Site, Vienna, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Wheeler CM, Harvey BM, Pichichero ME, Simon MW, Combs SP, Blatter MM, Marshall GS, Catteau G, Dobbelaere K, Descamps D, Dubin G, Schuind A. Immunogenicity and safety of human papillomavirus-16/18 AS04-adjuvanted vaccine coadministered with tetanus toxoid, reduced diphtheria toxoid, and acellular pertussis vaccine and/or meningococcal conjugate vaccine to healthy girls 11 to 18 years of age: results from a randomized open trial. Pediatr Infect Dis J. 2011 Dec;30(12):e225-34. doi: 10.1097/INF.0b013e31822d28df. PMID 21817954
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 107682 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107682 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 107682 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107682 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107682 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 107682 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cervarix + Boostrix/Menactra Group | Cervarix + Menactra/Boostrix Group | Cervarix + Boostrix + Menactra Group | Boostrix/Cervarix Group | Menactra/Cervarix Group | Cervarix Group
Started | 212 | 214 | 214 | 214 | 214 | 215
Completed | 197 | 195 | 202 | 199 | 196 | 204
Not Completed | 15 | 19 | 12 | 15 | 18 | 11
Not completed — Adverse Event | 0 | 2 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 9 | 5 | 5 | 4 | 6 | 2
Not completed — Lost to Follow-up | 6 | 11 | 7 | 8 | 9 | 6
Not completed — Other | 0 | 0 | 0 | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix + Boostrix/Menactra Group | Cervarix + Menactra/Boostrix Group | Cervarix + Boostrix + Menactra Group | Boostrix/Cervarix Group | Menactra/Cervarix Group | Cervarix Group | Total
Number analyzed (Participants) | 212 | 214 | 214 | 214 | 214 | 215 | 1283
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.5 (2.27) | 13.3 (2.28) | 13.5 (2.26) | 13.5 (2.33) | 13.3 (2.35) | 13.4 (2.34) | 13.4 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 212 | 214 | 214 | 214 | 214 | 215 | 1283
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-diphtheria Toxoid (Anti-D) and Anti-tetanus Toxoid (Anti-T) Antibody Concentrations Above 1.0 International Unit Per Milliliter (IU/mL)
Description: Anti-D and anti-T antibodies cut-off values assessed include 1.0 international unit per milliliter (IU/mL)
Time Frame: Before and one month after vaccination with Boostrix
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity, Month 1 and only for Cervarix + Boostrix/Menactra, Cervarix + Boostrix + Menactra and Boostrix/Cervarix groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix + Boostrix/Menactra Group | Cervarix + Menactra/Boostrix Group | Cervarix + Boostrix + Menactra Group | Boostrix/Cervarix Group | Menactra/Cervarix Group | Cervarix Group
Number analyzed (Participants) | 194 | 0 | 201 | 199 | 0 | 0
Participants
  Anti-D (Before vaccination): number analyzed (Participants) | 193 | 0 | 199 | 199 | 0 | 0
  Anti-D (Before vaccination) | 38 |  | 33 | 39 |  |
  Anti-D (1 month after vaccination) | 193 |  | 200 | 190 |  |
  Anti-T (Before vaccination): number analyzed (Participants) | 194 | 0 | 199 | 199 | 0 | 0
  Anti-T (Before vaccination) | 75 |  | 75 | 72 |  |
  Anti-T (1 month after vaccination) | 194 |  | 201 | 198 |  |

2. Primary Outcome: Concentration of Anti-pertussis Toxoid (Anti-PT), Anti-pertactin (Anti-PRN) and Anti-filamentous Hemagglutinin (Anti-FHA) Antibodies
Description: Concentrations given as Geometric Means Concentrations (GMCs)
Time Frame: Before and one month after vaccination with Boostrix
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity Month 1, and only for Cervarix + Boostrix/Menactra, Cervarix + Boostrix + Menactra and Boostrix/Cervarix groups.
Measure: Geometric Mean (95% Confidence Interval); unit: International Units per Milliliter
Arm/Group | Cervarix + Boostrix/Menactra Group | Cervarix + Menactra/Boostrix Group | Cervarix + Boostrix + Menactra Group | Boostrix/Cervarix Group | Menactra/Cervarix Group | Cervarix Group
Number analyzed (Participants) | 194 | 0 | 201 | 199 | 0 | 0
International Units per Milliliter
  Anti-PT (Before vaccination): number analyzed (Participants) | 194 | 0 | 196 | 198 | 0 | 0
  Anti-PT (Before vaccination) | 9.515 [8.078 to 11.207] |  | 10.356 [8.733 to 12.280] | 11.164 [9.319 to 13.375] |  |
  Anti-PT (1month after vaccination) | 74.682 [66.001 to 84.504] |  | 70.908 [61.763 to 81.408] | 78.807 [69.035 to 89.962] |  |
  Anti-FHA (Before vaccination): number analyzed (Participants) | 192 | 0 | 195 | 196 | 0 | 0
  Anti-FHA (Before vaccination) | 32.472 [27.019 to 39.026] |  | 37.671 [31.572 to 44.947] | 38.819 [32.467 to 46.413] |  |
  Anti-FHA (1month after vaccination) | 648.018 [577.051 to 727.714] |  | 544.665 [481.612 to 615.974] | 676.765 [596.493 to 767.840] |  |
  Anti-PRN (Before vaccination): number analyzed (Participants) | 193 | 0 | 199 | 199 | 0 | 0
  Anti-PRN (Before vaccination) | 12.978 [10.781 to 15.622] |  | 16.040 [13.479 to 19.087] | 15.871 [13.033 to 19.327] |  |
  Anti-PRN(1month after vaccination): number analyzed (Participants) | 194 | 0 | 199 | 198 | 0 | 0
  Anti-PRN(1month after vaccination) | 416.049 [345.557 to 500.921] |  | 323.205 [268.389 to 389.217] | 379.467 [311.050 to 462.933] |  |

3. Primary Outcome: Titer of Meningococcal Serogroup A (Anti-A), Meningococcal Serogroup C (Anti-C), Meningococcal Serogroup Y (Anti-Y) and Meningococcal Serogroup W-135 (Anti-W135) Antibodies
Description: Titers given as Geometric Mean Titers (GMTs)
Time Frame: Before and one month after vaccination with Menactra
Population: Analysis was performed on the According to Protocol (ATP) cohort for immunogenicity Month1 and only for Cervarix + Menactra/Boostrix, Cervarix + Boostrix + Menactra and Menactra/Cervarix groups.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cervarix + Boostrix/Menactra Group | Cervarix + Menactra/Boostrix Group | Cervarix + Boostrix + Menactra Group | Boostrix/Cervarix Group | Menactra/Cervarix Group | Cervarix Group
Number analyzed (Participants) | 0 | 200 | 200 | 0 | 203 | 0
Titer
  Anti-A (Before vaccination): number analyzed (Participants) | 0 | 180 | 179 | 0 | 184 | 0
  Anti-A (Before vaccination) |  | 898.650 [780.476 to 1034.717] | 829.508 [716.806 to 959.931] |  | 763.324 [648.325 to 898.721] |
  Anti-A (1month after vaccination): number analyzed (Participants) | 0 | 190 | 181 | 0 | 184 | 0
  Anti-A (1month after vaccination) |  | 7570.228 [6701.054 to 8556.140] | 6919.419 [6197.308 to 7725.670] |  | 8352.685 [7435.325 to 9383.226] |
  Anti-C (Before vaccination): number analyzed (Participants) | 0 | 184 | 190 | 0 | 182 | 0
  Anti-C (Before vaccination) |  | 37.738 [27.249 to 52.264] | 35.827 [26.004 to 49.360] |  | 30.696 [21.974 to 42.879] |
  Anti-C (1month after vaccination) |  | 2497.463 [1985.199 to 3141.912] | 2112.366 [1708.155 to 2612.228] |  | 2375.963 [1938.868 to 2911.595] |
  Anti-Y (Before vaccination): number analyzed (Participants) | 0 | 183 | 189 | 0 | 192 | 0
  Anti-Y (Before vaccination) |  | 87.356 [63.239 to 120.670] | 72.756 [52.881 to 100.101] |  | 110.911 [81.291 to 151.322] |
  Anti-Y (1month after vaccination) |  | 4787.556 [4079.870 to 5617.996] | 3947.330 [3292.007 to 4733.105] |  | 4335.380 [3688.566 to 5095.617] |
  Anti-W135 (Before vaccination): number analyzed (Participants) | 0 | 185 | 188 | 0 | 189 | 0
  Anti-W135 (Before vaccination) |  | 33.946 [24.902 to 46.274] | 28.750 [21.338 to 38.737] |  | 34.206 [25.374 to 46.111] |
  Anti-W135(1month after vaccination): number analyzed (Participants) | 0 | 200 | 200 | 0 | 201 | 0
  Anti-W135(1month after vaccination) |  | 4564.037 [3990.523 to 5219.977] | 3856.584 [3298.787 to 4508.700] |  | 5056.182 [4401.292 to 5808.516] |

4. Secondary Outcome: Number of Subjects With Anti-human Papilloma Virus 16 (Anti-HPV16) and Anti-human Papilloma Virus 18 (Anti-HPV18) Antibody Concentrations Above Pre-defined Cut-off Values
Description: Cut-off values assessed include 8 enzyme-linked immunosorbent assay units Per Milliliter (EL.U/mL) for anti-HPV16 antibodies and 7 EL.U/mL for anti-HPV18 antibodies.
Time Frame: Before vaccination (PRE), one month post Dose 2 (Mth2) and one and six months post Dose 3 (Mth 7 and Mth 12)
Population: Analysis was performed on the According to Protocol (ATP) cohort for immunogenicity at Month 12/13
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix + Boostrix/Menactra Group | Cervarix + Menactra/Boostrix Group | Cervarix + Boostrix + Menactra Group | Boostrix/Cervarix Group | Menactra/Cervarix Group | Cervarix Group
Number analyzed (Participants) | 163 | 158 | 165 | 156 | 147 | 166
Participants
  Anti-HPV16 PRE: number analyzed (Participants) | 163 | 158 | 164 | 156 | 146 | 166
  Anti-HPV16 PRE | 19 | 8 | 9 | 5 | 11 | 11
  Anti-HPV16 Mth2: number analyzed (Participants) | 163 | 158 | 163 | 156 | 145 | 166
  Anti-HPV16 Mth2 | 163 | 158 | 163 | 156 | 145 | 166
  Anti-HPV16 Mth7: number analyzed (Participants) | 161 | 158 | 164 | 156 | 142 | 164
  Anti-HPV16 Mth7 | 161 | 158 | 164 | 156 | 142 | 164
  Anti-HPV16 Mth12: number analyzed (Participants) | 163 | 158 | 164 | 156 | 146 | 166
  Anti-HPV16 Mth12 | 163 | 158 | 164 | 156 | 146 | 166
  Anti-HPV18 PRE: number analyzed (Participants) | 163 | 157 | 165 | 152 | 147 | 165
  Anti-HPV18 PRE | 14 | 10 | 13 | 8 | 6 | 11
  Anti-HPV18 Mth2: number analyzed (Participants) | 163 | 157 | 164 | 152 | 146 | 165
  Anti-HPV18 Mth2 | 163 | 157 | 164 | 152 | 146 | 165
  Anti-HPV18 Mth7: number analyzed (Participants) | 161 | 157 | 165 | 152 | 143 | 163
  Anti-HPV18 Mth7 | 161 | 157 | 165 | 152 | 143 | 163
  Anti-HPV18 Mth12: number analyzed (Participants) | 163 | 157 | 165 | 152 | 147 | 165
  Anti-HPV18 Mth12 | 163 | 157 | 165 | 152 | 147 | 165

5. Secondary Outcome: Number of Subjects With Anti-diphtheria Toxoid (Anti-D) and Anti-tetanus Toxoid (Anti-T) Antibody Concentrations Above 0.1 International Unit Per Milliliter (IU/mL)
Description: Anti-D and anti-T antibodies cut-off values assessed include 0.1 international unit per milliliter (IU/mL)
Time Frame: Before and one month after vaccination with Boostrix
Population: Analysis was performed on the According to Protocol (ATP) cohort for immunogenicity Month 1, and only for Cervarix + Boostrix/Menactra, Cervarix + Boostrix + Menactra and Boostrix/Cervarix groups
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix + Boostrix/Menactra Group | Cervarix + Menactra/Boostrix Group | Cervarix + Boostrix + Menactra Group | Boostrix/Cervarix Group | Menactra/Cervarix Group | Cervarix Group
Number analyzed (Participants) | 194 | 0 | 201 | 199 | 0 | 0
Participants
  Anti-D (Before vaccination): number analyzed (Participants) | 193 | 0 | 199 | 199 | 0 | 0
  Anti-D (Before vaccination) | 170 |  | 181 | 167 |  |
  Anti-D (1month after vaccination) | 194 |  | 201 | 199 |  |
  Anti-T (Before vaccination): number analyzed (Participants) | 194 | 0 | 199 | 199 | 0 | 0
  Anti-T (Before vaccination) | 188 |  | 199 | 195 |  |
  Anti-T (1month after vaccination) | 194 |  | 201 | 199 |  |

6. Secondary Outcome: Concentration of Anti-D and Anti-T Antibodies
Description: Concentrations given as Geometric Mean Concentrations (GMCs)
Time Frame: Before and one month after vaccination with Boostrix
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: International Unit per Milliliter
Arm/Group | Cervarix + Boostrix/Menactra Group | Cervarix + Menactra/Boostrix Group | Cervarix + Boostrix + Menactra Group | Boostrix/Cervarix Group | Menactra/Cervarix Group | Cervarix Group
Number analyzed (Participants) | 194 | 0 | 201 | 199 | 0 | 0
International Unit per Milliliter
  Anti-D (Before vaccination): number analyzed (Participants) | 193 | 0 | 199 | 199 | 0 | 0
  Anti-D (Before vaccination) | 0.362 [0.305 to 0.431] |  | 0.368 [0.315 to 0.430] | 0.331 [0.280 to 0.390] |  |
  Anti-D (1month after vaccination) | 8.928 [7.821 to 10.192] |  | 27.438 [24.297 to 30.984] | 7.527 [6.492 to 8.727] |  |
  Anti-T (Before vaccination): number analyzed (Participants) | 194 | 0 | 199 | 199 | 0 | 0
  Anti-T (Before vaccination) | 0.811 [0.686 to 0.960] |  | 0.895 [0.765 to 1.046] | 0.700 [0.602 to 0.814] |  |
  Anti-T (1month after vaccination) | 15.584 [13.923 to 17.443] |  | 12.415 [11.184 to 13.781] | 14.524 [12.814 to 16.462] |  |

7. Secondary Outcome: Number of Subjects With Booster Response for Anti-D and Anti-T
Description: Booster responses for anti-D and anti-T defined as:
  * For initially seronegative subjects (pre-vaccination titer below cut-off: < 0.1 IU/mL): antibody titer at least 4 times the cut-off (post-vaccination titer ≥ 0.4 IU/mL)
  * For initially seropositive subjects (pre-vaccination titer above 0.1 IU/mL): an increase in antibody titer of at least 4 times the pre-vaccination titer
Time Frame: One month after vaccination with Boostrix
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix + Boostrix/Menactra Group | Cervarix + Menactra/Boostrix Group | Cervarix + Boostrix + Menactra Group | Boostrix/Cervarix Group | Menactra/Cervarix Group | Cervarix Group
Number analyzed (Participants) | 194 | 0 | 199 | 199 | 0 | 0
Participants
  Anti-D: number analyzed (Participants) | 193 | 0 | 199 | 199 | 0 | 0
  Anti-D | 175 |  | 196 | 182 |  |
  Anti-T | 157 |  | 162 | 168 |  |

8. Secondary Outcome: Number of Subjects With Booster Response for Anti-PT, Anti-FHA and Anti-PRN
Description: Booster responses defined as:
  * For initially seronegative subjects (pre-vaccination titer below cut-off: < 5 EL.U/mL): antibody titers at least 4 times the cut-off,
  * For initially seropositive subjects with pre-vaccination titer above 5 EL.U/mL and < 20 EL.U/mL: an increase in antibody titers of at least 4 times the pre-vaccination titer,
  * For initially seropositive subjects with pre-vaccination titer ≥ 20 EL.U/mL: an increase in antibody titers of at least two times the pre-vaccination titer
Time Frame: One month after vaccination with Boostrix
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity Month 1, and only for Cervarix + Boostrix/Menactra, Cervarix + Boostrix + Menactra and Boostrix + Cervarix groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix + Boostrix/Menactra Group | Cervarix + Menactra/Boostrix Group | Cervarix + Boostrix + Menactra Group | Boostrix/Cervarix Group | Menactra/Cervarix Group | Cervarix Group
Number analyzed (Participants) | 194 | 0 | 197 | 198 | 0 | 0
Participants
  Anti-PT: number analyzed (Participants) | 194 | 0 | 196 | 198 | 0 | 0
  Anti-PT | 138 |  | 116 | 133 |  |
  Anti-FHA: number analyzed (Participants) | 192 | 0 | 195 | 196 | 0 | 0
  Anti-FHA | 167 |  | 163 | 165 |  |
  Anti-PRN: number analyzed (Participants) | 193 | 0 | 197 | 198 | 0 | 0
  Anti-PRN | 183 |  | 180 | 177 |  |

9. Secondary Outcome: Number of Subjects With Anti-A, Anti-C, Anti-Y and Anti-W135 Vaccine Response
Description: Vaccine responses for anti-A, C, Y and W-135 defined as:
  * For initially seronegative subjects (pre-vaccination titer below cut-off of 8): antibody titers at least 4 times the cut-off (post vaccination titer ≥ 32)
  * For initially seropositive subjects (pre-vaccination titer above 8): antibody titers at least 4 times the pre-vaccination antibody titer
Time Frame: One month after vaccination with Menactra
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity Month 1, and only for Cervarix + Menactra/Boostrix, Cervarix + Boostrix + Menactra and Menactra/Cervarix groups
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix + Boostrix/Menactra Group | Cervarix + Menactra/Boostrix Group | Cervarix + Boostrix + Menactra Group | Boostrix/Cervarix Group | Menactra/Cervarix Group | Cervarix Group
Number analyzed (Participants) | 0 | 185 | 189 | 0 | 192 | 0
Participants
  Anti-A: number analyzed (Participants) | 0 | 170 | 160 | 0 | 167 | 0
  Anti-A |  | 127 | 112 |  | 139 |
  Anti-C: number analyzed (Participants) | 0 | 184 | 189 | 0 | 182 | 0
  Anti-C |  | 162 | 163 |  | 161 |
  Anti-Y: number analyzed (Participants) | 0 | 183 | 188 | 0 | 192 | 0
  Anti-Y |  | 169 | 166 |  | 171 |
  Anti-W135: number analyzed (Participants) | 0 | 185 | 187 | 0 | 187 | 0
  Anti-W135 |  | 176 | 183 |  | 181 |

10. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling.
Time Frame: During the 7-day period following each vaccination
Population: Analysis was performed on the Total Vaccinated cohort including all vaccinated subjects receiving one dose at least
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix + Boostrix/Menactra Group | Cervarix + Menactra/Boostrix Group | Cervarix + Boostrix + Menactra Group | Boostrix/Cervarix Group | Menactra/Cervarix Group | Cervarix Group
Number analyzed (Participants) | 209 | 208 | 209 | 211 | 209 | 210
Participants
  Pain | 197 | 204 | 204 | 203 | 193 | 201
  Redness | 97 | 93 | 103 | 103 | 99 | 93
  Swelling | 94 | 90 | 102 | 100 | 74 | 86

11. Secondary Outcome: Number of Subjects Reporting Solicited General Symptoms
Description: Solicited general symptoms assessed include Arthralgia, fatigue, fever, gastrointestinal, headache, myalgia, rash and urticaria
Time Frame: During the 7-day period following each vaccination
Population: Analysis was performed on the Total Vaccinated cohort including all vaccinated subjects receiving one dose at least
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix + Boostrix/Menactra Group | Cervarix + Menactra/Boostrix Group | Cervarix + Boostrix + Menactra Group | Boostrix/Cervarix Group | Menactra/Cervarix Group | Cervarix Group
Number analyzed (Participants) | 209 | 208 | 210 | 211 | 209 | 210
Participants
  Arthralgia | 37 | 42 | 34 | 48 | 33 | 47
  Fatigue | 94 | 100 | 111 | 118 | 99 | 98
  Fever | 31 | 32 | 24 | 28 | 35 | 23
  Gastrointestinal | 59 | 62 | 70 | 65 | 65 | 69
  Headache | 107 | 118 | 124 | 133 | 122 | 112
  Myalgia | 80 | 89 | 101 | 96 | 66 | 89
  Rash | 11 | 12 | 19 | 15 | 13 | 13
  Urticaria | 7 | 5 | 12 | 7 | 4 | 6

12. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: Unsolicited adverse event = Any adverse event (AE) reported in addition to those solicited during the clinical study. Also any "solicited" symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event.
Time Frame: During the 30-day period following each vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix + Boostrix/Menactra Group | Cervarix + Menactra/Boostrix Group | Cervarix + Boostrix + Menactra Group | Boostrix/Cervarix Group | Menactra/Cervarix Group | Cervarix Group
Number analyzed (Participants) | 212 | 214 | 214 | 214 | 214 | 215
Participants | 108 | 121 | 119 | 122 | 127 | 118

13. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events
Description: Serious adverse events assessed include medical occurrences that results in death, is life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: During the active phase of the study (up to Month 7 or Month 8) and throughout the entire study (up to Month 12 or Month 13)
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix + Boostrix/Menactra Group | Cervarix + Menactra/Boostrix Group | Cervarix + Boostrix + Menactra Group | Boostrix/Cervarix Group | Menactra/Cervarix Group | Cervarix Group
Number analyzed (Participants) | 212 | 214 | 214 | 214 | 214 | 215
Participants
  During the active phase | 0 | 2 | 3 | 0 | 5 | 4
  During the entire study | 1 | 3 | 4 | 0 | 7 | 4

14. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events as New Onset Chronic Diseases (NOCDs)
Description: NOCDs assessed include e.g. autoimmune disorders, asthma, type I diabetes
Time Frame: During the active phase of the study (up to Month 7 or Month 8) and throughout the entire study period (up to Month 12 or Month 13)
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix + Boostrix/Menactra Group | Cervarix + Menactra/Boostrix Group | Cervarix + Boostrix + Menactra Group | Boostrix/Cervarix Group | Menactra/Cervarix Group | Cervarix Group
Number analyzed (Participants) | 212 | 214 | 214 | 214 | 214 | 215
Participants
  During the active phase | 3 | 6 | 6 | 5 | 11 | 6
  During the entire study | 3 | 6 | 6 | 6 | 12 | 6

15. Secondary Outcome: Number of Subjects Reporting Medically Significant Adverse Events (AEs)
Description: Medically significant AEs assessed include AEs prompting emergency room or physician visits that are not related to common diseases or SAEs that are not related to common diseases.
Time Frame: During the active phase (up to Month 7 or Month 8) and throughout the entire study (up to Month 12 or Month 13)
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix + Boostrix/Menactra Group | Cervarix + Menactra/Boostrix Group | Cervarix + Boostrix + Menactra Group | Boostrix/Cervarix Group | Menactra/Cervarix Group | Cervarix Group
Number analyzed (Participants) | 212 | 214 | 214 | 214 | 214 | 215
Participants
  During the active phase | 40 | 43 | 51 | 56 | 62 | 59
  During the entire study | 43 | 46 | 54 | 59 | 64 | 64

ADVERSE EVENTS:
Arm/Group | Cervarix + Boostrix/Menactra Group | Cervarix + Menactra/Boostrix Group | Cervarix + Boostrix + Menactra Group | Boostrix/Cervarix Group | Menactra/Cervarix Group | Cervarix Group
Serious Adverse Events (participants affected / at risk) | 1 | 3 | 4 | 0 | 7 | 4
Other Adverse Events (participants affected / at risk) | 202/212 | 207/214 | 205/214 | 208/214 | 202/214 | 203/215
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Cervarix + Boostrix/Menactra Group | Cervarix + Menactra/Boostrix Group | Cervarix + Boostrix + Menactra Group | Boostrix/Cervarix Group | Menactra/Cervarix Group | Cervarix Group
Appendicitis (Infections and infestations) | 0/212 | 1/214 | 0/214 | 0/214 | 2/214 | 0/215
Abdominal pain (Gastrointestinal disorders) | 0/212 | 0/214 | 0/214 | 0/214 | 1/214 | 0/215
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 0/212 | 0/214 | 0/214 | 0/214 | 1/214 | 0/215
Adjustment disorder (Psychiatric disorders) | 0/212 | 0/214 | 0/214 | 0/214 | 0/214 | 1/215
Bipolar disorder (Psychiatric disorders) | 0/212 | 0/214 | 0/214 | 0/214 | 1/214 | 0/215
Dehydration (Metabolism and nutrition disorders) | 0/212 | 0/214 | 0/214 | 0/214 | 0/214 | 1/215
Drug hypersensitivity (Immune system disorders) | 0/212 | 0/214 | 0/214 | 0/214 | 1/214 | 0/215
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0/212 | 0/214 | 0/214 | 0/214 | 0/214 | 1/215
Gastroenteritis viral (Infections and infestations) | 0/212 | 0/214 | 0/214 | 0/214 | 0/214 | 1/215
Hyphaema (Eye disorders) | 0/212 | 0/214 | 1/214 | 0/214 | 0/214 | 0/215
Ligament rupture (Injury, poisoning and procedural complications) | 0/212 | 0/214 | 1/214 | 0/214 | 0/214 | 0/215
Neutropenia (Blood and lymphatic system disorders) | 0/212 | 0/214 | 0/214 | 0/214 | 1/214 | 0/215
Pyrexia (General disorders) | 0/212 | 0/214 | 0/214 | 0/214 | 1/214 | 0/215
Rash pruritic (Skin and subcutaneous tissue disorders) | 0/212 | 0/214 | 0/214 | 0/214 | 1/214 | 0/215
Staphylococcal infection (Infections and infestations) | 0/212 | 0/214 | 0/214 | 0/214 | 1/214 | 0/215
Stevens-johnson syndrome (Skin and subcutaneous tissue disorders) | 0/212 | 1/214 | 0/214 | 0/214 | 0/214 | 0/215
Urinary tract infection (Infections and infestations) | 0/212 | 0/214 | 0/214 | 0/214 | 1/214 | 0/215
Viral infection (Infections and infestations) | 0/212 | 0/214 | 1/214 | 0/214 | 0/214 | 0/215
Conversion disorder (Psychiatric disorders) | 0/212 | 0/214 | 1/214 | 0/214 | 0/214 | 0/215
Depression (Psychiatric disorders) | 0/212 | 1/214 | 0/214 | 0/214 | 0/214 | 0/215
Facial palsy (Nervous system disorders) | 1/212 | 0/214 | 0/214 | 0/214 | 0/214 | 0/215
Proctitis (Gastrointestinal disorders) | 0/212 | 0/214 | 0/214 | 0/214 | 1/214 | 0/215
Suicidal ideation (Psychiatric disorders) | 0/212 | 1/214 | 0/214 | 0/214 | 0/214 | 0/215
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix + Boostrix/Menactra Group (N=212) | Cervarix + Menactra/Boostrix Group (N=214) | Cervarix + Boostrix + Menactra Group (N=214) | Boostrix/Cervarix Group (N=214) | Menactra/Cervarix Group (N=214) | Cervarix Group (N=215)
Pain (General disorders) | 197 | 204 | 204 | 203 | 193 | 201
Redness (General disorders) | 97 | 93 | 103 | 103 | 99 | 93
Swelling (General disorders) | 94 | 90 | 102 | 100 | 74 | 86
Arthralgia (General disorders) | 37 | 42 | 34 | 48 | 33 | 47
Fatigue (General disorders) | 94 | 100 | 111 | 118 | 99 | 98
Fever (General disorders) | 31 | 32 | 24 | 28 | 35 | 23
Gastrointestinal (General disorders) | 59 | 62 | 70 | 65 | 65 | 69
Headache (General disorders) | 107 | 118 | 124 | 133 | 122 | 112
Myalgia (General disorders) | 80 | 89 | 101 | 96 | 66 | 89
Rash (General disorders) | 11 | 12 | 19 | 15 | 13 | 13
Urticaria (General disorders) | 7 | 5 | 12 | 7 | 4 | 6
Injection site haematoma (General disorders) | 37 | 35 | 29 | 31 | 22 | 17
Headache (Nervous system disorders) | 13 | 16 | 13 | 13 | 21 | 18
Nasopharynigitis (Infections and infestations) | 11 | 13 | 13 | 10 | 16 | 18
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 8 | 0 | 10 | 13 | 15
Upper respiratory tract infection (Infections and infestations) | 0 | 10 | 12 | 14 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 9 | 0 | 13 | 10 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 10 | 0 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 11 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.